CLINICAL TRIAL: NCT06468111
Title: Efficacy Study of Dog-Assisted Therapy in Children During Blood or Dental Extraction: Extra-can Project
Brief Title: Dog-Assisted Therapy in Children During Blood or Dental Extraction.
Acronym: Extra-can
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Public Health Service of Cataluña (Other)
Responsible Party: Principal Investigator, Esther Rodrigo Claverol, Graduate in Medicine, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DMP ID: 2163
Record Dates: First submitted 2024-06-09; First posted 2024-06-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Emotional Stress
Keywords: Animal-assisted Intervention; Children; Primary Healthcare Centre; Venipuncture; Dental fear; Distraction emotional support animals
MeSH Terms: conditions — Stress, Psychological | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, two-arm clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group underwent a blood and dental extraction will be performed according to the usual protocol of the health center.
  Interventions: Behavioral: Animal Assisted Therapy
- experimental group (Experimental): The experimental group underwent a blood and dental extraction will be performed according to the usual protocol of the health center, the same as control group, and in addition dog-assisted therapy will be performed.
  Intervention (with the additional assistance of the therapy dog). Includes AAT with 10 minutes of pre-procedure interaction with the therapy dog, extraction performed with the therapy dog, and 5 minutes of post-procedure interaction.
  Interventions: Behavioral: Animal Assisted Therapy

INTERVENTIONS:
Behavioral: Animal Assisted Therapy — Blood and dental extraction will be performed according to the usual protocol of the health center in both groups; with the additional assistance of the therapy dog in experimental group.
  Other Names: Dog Assisted Therapy

SUMMARY:
The purpose of the present study is to evaluate the efficacy of Animal Assisted Therapy (AAT) during blood extraction or dental procedures in a Primary Care Pediatric Service. Determine the improvement in facilitating the task of venipuncture or dental extraction for nursing or dental professionals. Estimate the reduction in the child's emotional stress during these procedures with the support of a therapy dog. Evaluate the emotional stress in the accompanying family member. These objectives will be accomplished through a randomized open label two-arm controlled study of AAT for children who need a blood or dental extraction.

DETAILED DESCRIPTION:
INTRODUCTION: Venous puncture for routine blood sampling can be distressing for many children, leading to heightened anxiety both before and during the procedure. Dental anxiety affects around 9% of European children and adolescents, potentially persisting into adulthood and resulting in dental avoidance behaviors. Animal-assisted therapy (AAT) is viewed as a distraction technique that could play a vital role in managing pain and distress for children. AAT is a planned, structured therapeutic intervention with specific goals, facilitated by healthcare professionals.

OBJECTIVES: Evaluate the efficacy of AAT during blood or dental extraction in a Primary Care Pediatric Service. Determine the improvement in facilitating the task of venipuncture or dental extraction for nursing or dental professionals. Estimate the reduction in the child's emotional stress during these procedures with the support of a therapy dog. Evaluate the emotional stress in the accompanying family member.

METHODOLOGY: Randomized two-arm clinical trial (control group and intervention group) involving children aged 3 to 8 requiring blood analysis or dental extraction in a Primary Health Care Center. Patients will be randomly assigned to the control and intervention groups. Sample size calculations suggest 60 patients in each group to detect statistically significant differences. The control group follows standard protocols, while the intervention group includes AAT with 10 minutes of pre-procedure interaction with the therapy dog, extraction performed with the therapy dog, and 5 minutes of post-procedure interaction. Personnel includes nurses or dentists, a pediatrician, and an AAT technician. Response variables include various scales measuring anxiety and distress, while control variables encompass age, gender, pathologies, extraction type, and pet ownership.

EXPECTED RESULTS: The implementation of AAT as an emotional support intervention, utilizing a therapy dog for distraction, is anticipated to improve symptomatology in the intervention group by reducing fear and anxiety post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 12 years old.
* Need a blood or dental extraction.
* Willing to participate in the study on a voluntary basis.
* Delivery of the information sheet and signature the informed consent.

Exclusion Criteria:

* If in the initial interview they declared having allergy or fear of dogs.
* Have aggression disorder towards dogs.
* Not want to participate in the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Observation Scale of Behavioral Distress (OSBD) registered at baseline, during and immediately after the intervention | This scale registered behaviors in continuous 15-second intervals at baseline, during and immediately after the intervention
  Is an instrument for measuring children's distress during painful medical procedures, assessed by an external observer. It is a 4-point Likert-type scale instrument (where the numerical values are weighted from 0 (not at all) to 3 (very much)) that evaluates 11 different behaviors

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory Questionnaire (STAI) registered at baseline and immediately after the intervention | This questionnaire will be administered at baseline and immediately after the intervention, post-extraction.
  Is a self-administered questionnaire that assesses the levels of clinical anxiety (both trait anxiety ("most of the time") and state anxiety ("at the present moment")). The total score on each of the subscales ranges from 0 to 60 points.
Wong-Baker Faces Scale registered at baseline and immediately after the intervention | This scale will be administered at baseline and immediately after the intervention, post-extraction.
  Is a tool that uses a combination of faces, numbers, and words to help a person effectively communicate the severity of their physical pain. A 0 point 'happy face' represents the absence or lack of pain. A 10 point 'crying face' represents the worst possible or most excruciating pain. All the faces in between represent a scoring of 2, 4, 6, or 8, respectively, based on the pain severity facial image chosen.

OTHER OUTCOMES:
Evaluation questionnaire for health professionals administered immediately after the intervention | This questionnaire will be administered immediately after the intervention, post-extraction
  This is a questionnaire that will be completed by the professionals (nursing or dentist) at the end of the intervention. Using a Likert scale from 0 to 10 (0= Not at all and 10= A lot). It contains the following questions:
  * Did you find it stressful to do the extraction? (CG+EG)
  * How relaxed you have seen the child? (CG+EG)
  * How calm have you seen the parents? (CG+EG)
  * Did the presence of the dog make the extraction easier? (EG)
  * Do you consider that the dog reduces the risk of accidents during extraction? (EG)
  * Has the presence of the dog interfered with your work? (EG)
Parent satisfaction questionnaire administered immediately after the intervention | This questionnaire will be administered immediately after the intervention, post-extraction
  The following questions will be asked in writing and answered by parents.Using a Likert scale from 0 to 10 (0= Not at all and 10= A lot). It contains the following questions:
  * Have you experienced this procedure (extraction) in a stressful way? (CG+EG)
  * How relaxed have you seen the child? (CG+EG)
  * In terms of satisfaction, how would you rate this procedure? (CG+EG)
  * Has the presence of the dog made the child feel calmer? (EG)
  * Has the presence of the dog made you feel calmer? (EG)
  * Do you think that the child has experienced the extraction as a less aggressive activity because of the presence of the dog? (EG)
  * Would you recommend this experience to other parents to do with their children? (EG)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ortega Bravo, PhD, Study Director — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Centre d'Atenció Primària Primer de Maig, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No